CLINICAL TRIAL: NCT02520570
Title: Post-market Safety Reassessment of Ulinastatin for Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Techpool Bio-Pharma Co., Ltd. (Industry)
Collaborators: Center for ADR Monitoring of Guangdong (Unknown)
Responsible Party: Sponsor
Other Study IDs: 002/20140709
Record Dates: First submitted 2015-07-30; First posted 2015-08-13 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Adverse Reaction to Drug
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — urinastatin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- general department: Patients using ulinastatin in department beyond ICU would be labelled as general department group.
  Interventions: Drug: ulinastatin
- ICU: Patients using ulinastatin in ICU would be labelled as ICU group.
  Interventions: Drug: ulinastatin

INTERVENTIONS:
Drug: ulinastatin — We wouldn't intervene the doctors how to treat with the patients or how to use the drug, we just observe the react of patients after treated with ulinastatin.
  Other Names: UTI; urinary trypsin inhibitor; bikunin

SUMMARY:
1. Investigate the application of ulinastatin(UTI) in real practice clinic.(eg:population character, usage and dosage, course of treatment,etc )
2. Analysis the incidence of adverse drug reactions /adverse events of ulinastatin, collect the main clinical manifestations, treatment, outcome, influence factors; provide evidence for improving the recommended medication plan of ulinastatin.
3. Evaluate the safety of ulinastatin , obtain scientific conclusion , and provide evidence for appropriate medication to administration department of health authority.

DETAILED DESCRIPTION:
In order to find out the application of ulinastatin in real practice clinic , identify the high risk group for adverse event/adverse drug reaction and calculate the adverse event/adverse drug reaction incidence rate, a large sample size clinical trial has been designed. This trial is an observational study. The investigators would screen several hospitals from different provinces and prospectively collect the main clinical manifestations,treatment, outcome, influence factors about patients using ulinastatin either in general clinical departments or in ICU. This study would be expected to provide evidence for appropriate medication to administration department of health authority.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulinastatin treated

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with ulinastatin treated
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | participants will be followed for the duration of using ulinastatin, an expected average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, doctor, Principal Investigator — Center for Adverse Drug Reaction Monitoring of Guangdong
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided